CLINICAL TRIAL: NCT02742506
Title: Beneficial Effects of Music on Cognition and Consciousness Level
Acronym: MUSICOREVEIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2012.750; 2012-A01025-38 (Other: ID-RCB)
Record Dates: First submitted 2016-04-07; First posted 2016-04-19 (Estimated); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Coma
Keywords: Brain-damaged; Disorders of consciousness; Post-coma; consciousness; coma; vegetative state; minimally conscious state; music; P300
MeSH Terms: conditions — Coma; Consciousness Disorders; Persistent Vegetative State

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (2):
- Brain-damaged patients (Experimental): Electroencephalography (EEG) will be performed in patients in coma, in a vegetative state or in a minimally conscious state to assess the P300 response after different auditive stimulations
  Interventions: Other: Electroencephalography (EEG)
- Healthy volunteers (Active Comparator): Electroencephalography (EEG) will be performed in healthy participants to assess the P300 response and medial prefrontal cortex activity after different auditive stimulations
  Interventions: Other: Electroencephalography (EEG)

INTERVENTIONS:
Other: Electroencephalography (EEG) — EEG will be performed to assess brain activity in response to sounds of different nature, including music and the given name of the registered person

SUMMARY:
Exposure to music improves cognitive function in 'healthy' participants and in brain-damaged patients. However, it is still difficult to understand what precisely in music causes a positive effect : are they emotional components, familiarity or preference which improve cognition or is there any specific effect of music? Moreover, it is not yet possible to characterize the neural and functional links between the brain systems solicited by music and those associated with other cognitive functions enhanced by music.

Finally, researches on brain-damaged patients have not exploited the potential effect of music on the level of alert and perceptual awareness, while this type of stimulation could be a valuable tool to improve cognition in patients with a disturbance of consciousness and alertness.

The main objective is to describe the impact of music on the brain's response to self-referential or neutral stimuli in brain-damaged patients with persistent consciousness disorder after a coma and in healthy participants.

ELIGIBILITY:
Brain-damaged patients :

Inclusion Criteria:

* Disorders of consciousness (Traumatic brain injury, stroke or anoxic encephalopathy)
* Coma diagnosis (Plum and Posner, 1966), vegetative state (Task Force, 1994) or minimally conscious state (Giacino, Ashwal et al. 2002)
* Lack of autonomic crisis since one week minimum
* Medical condition considered stable
* Patients who do not present hearing loss. Peaks I and II of Brainstem Auditory Evoked Potentials (BAEP) will be normal.

Exclusion Criteria:

* Hearing Problem
* Uncontrolled Epilepsy
* Autonomic crises
* Medical unstable state
* Pregnant or likely to be (interrogation data) or breastfeeding woman

Healthy participants :

Inclusion Criteria:

* Subjects with normal hearing
* Absence of neurological disorder
* Subjects able to understand the experimental instructions

Exclusion Criteria:

* Hearing problems and / or hearing loss higher than 30 decibels Hearing Level (dB HL) at a frequency band from 250 to 8000 Hz
* Neurological disorders
* Pregnant or likely to be (interrogation data) or breastfeeding woman

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2013-06-25 (Actual); Primary Completion 2019-10-23 (Actual); Study Completion 2019-10-23 (Actual)

PRIMARY OUTCOMES:
P300 response in brain-damaged patients | 24 hours after inclusion
  Improvement of the P300 response (increase in amplitude and / or a decrease in latency) to the first name pronunciation will be assessed in patients in coma, in a vegetative state or in a minimally conscious state, when it is preceded by a favorite or familiar sound (music, language, environmental noise) and / or a positive emotional connotation, compared to a control condition (unfamiliar sound and / or neutral emotional connotation). This improvement in brain response will be the sign of a more efficient categorization of patient's own name.

SECONDARY OUTCOMES:
P300 response in healthy volunteers | 24 hours after inclusion
  Improvement of the P300 response (increase in amplitude and / or a decrease in latency) to a self-referential stimulation (eg first name pronunciation) compared to a non-self-referential stimulation (eg other name) will be assessed in healthy participants when it is preceded by a favorite or familiar sound (music, language, environmental noise) and / or a positive emotional connotation, compared to a control condition (sound unfamiliar and / or neutral emotional connotation)
P300 response in brain-damaged patients | 24 hours after inclusion
  Increase of the P300 response (increase in amplitude and / or a decrease in latency) to a self-referential stimulation (e.g. name pronunciation) will be assessed when the patient is awake (according to EEG measures and / or eye opening) compared to when the patient is asleep (according to EEG measures and / or eye closure).
Medial prefrontal cortex activity level in healthy volunteers | 24 hours after inclusion
  Increase of the level of activity measured in the medial prefrontal cortex will be assessed in healthy participants after a favorite or familiar sound (music, language, environmental noise) and / or a positive emotional connotation, compared to a control condition (unfamiliar sound and / or neutral emotional connotation).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon - Hôpital Neurologique Pierre Wertheimer - Service de Médecine Physique et Réadaptation, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Corneyllie A, Perrin F, Heine L. Sharing an Open Stimulation System for Auditory EEG Experiments Using Python, Raspberry Pi, and HifiBerry. eNeuro. 2021 Aug 25;8(4):ENEURO.0524-20.2021. doi: 10.1523/ENEURO.0524-20.2021. Print 2021 Jul-Aug. PMID 34301720
- [Background] Heine L, Corneyllie A, Gobert F, Luaute J, Lavandier M, Perrin F. Virtually spatialized sounds enhance auditory processing in healthy participants and patients with a disorder of consciousness. Sci Rep. 2021 Jul 1;11(1):13702. doi: 10.1038/s41598-021-93151-6. PMID 34211035
- [Background] Castro M, Tillmann B, Luaute J, Corneyllie A, Dailler F, Andre-Obadia N, Perrin F. Boosting Cognition With Music in Patients With Disorders of Consciousness. Neurorehabil Neural Repair. 2015 Sep;29(8):734-42. doi: 10.1177/1545968314565464. Epub 2015 Feb 3. PMID 25650390